CLINICAL TRIAL: NCT02240004
Title: Removal of Uremic Toxins and Improvement of Chronic Inflammation With HFR in Comparison With "On-Line" Hemodiafiltration and High Flux Hemodialysis.
Brief Title: Hemo Filtration Reinfusion (HFR) Clearance Efficiency Towards P-bound Toxins and Effects on Inflammatory and Endothelial Damage Markers
Acronym: SUPREMO
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Alejandro Martin-Malo, MD, Hospital Universitario Reina Sofia de Cordoba
Other Study IDs: CRB2014
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SUPRA HFR — usual dialytic prescription for duration, frequency, acid buffer and anticoagulation regimen

SUMMARY:
The aim of this study is to compare purification efficiency of HFR in terms of clearance of protein-bound toxins and the effects on markers of inflammation and endothelial damage, in comparison to HF-HD and OL-HDF.

DETAILED DESCRIPTION:
Protein-bound uremic toxins are poorly removed by current dialysis techniques because of their size, which is larger than the pore size of dialysis membranes available in the market. These protein-bound uremic toxins have emerged as important risk factors for progression of CKD, as well as for cardiovascular disease. Several studies have demonstrated that protein-bound uremic toxins induce vascular inflammation, endothelial dysfunction and vascular calcification.

In dialysis patients, serum concentrations of p-cresyl sulphate and indoxyl sulphate are approximately 17 and 54 times higher, respectively, than in healthy subjects. Because these toxins are bound to proteins, only a 30% or less is removed efficiently by hemodialysis. Traditional renal replacement therapies depend upon diffusion and convection for solute clearances and the use of an adsorbent in combination with dialysis membranes may be a new therapeutic option to increase removal rate of these uremic protein-bound toxins.

HFR technique uses a dual dialyzer with a resin between chambers. The first chamber is a high-flux membrane where convective process takes place. The ultrafiltrate obtained from this first chamber passes through the cartridge and is reinfused before the second chamber, a low-flux membrane, where diffusive process is performed.

In HFR, adsorption and haemodiafiltration are attached, using ultrafiltrate as a replacement fluid and being capable of theoretically removing most medium and high molecular weight uremic toxins. A potential benefit has been regarded for toxicity, biocompatibility, tolerance, and preservation of essential elements such as albumin, vitamins, amino acids or growth factors. An improvement on oxidative stress has also been described in HFR.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients on hemodialysis for al least 3 month
* older than 18 year old
* dialyzed at least for two months with a high-flux membrane permeability
* arteriovenous fistula with high blood flow (> 350 ml / min)

Exclusion Criteria:

* active neoplasia
* positive viral markers (HBsAg, anti-HCV and HIV),
* clinical signs of active infection and/or inflammation,
* albumin < 3.5 g/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing dialysis three times week
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory status: (CD14+ CD16+, CD14++ CD16+, cytokines levels) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- HU Reina Sofia, Córdoba, Spain